CLINICAL TRIAL: NCT00361465
Title: Characterization of Dystonia and Influence of Cognitive-attentional Factors
Brief Title: DYSCAR: Characterization of Dystonia
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Pierre POLLAK-Professor, University Joseph Fourier, INSERM U318, Grenoble University Hospital
Other Study IDs: 0610
Record Dates: First submitted 2006-08-07; First posted 2006-08-08 (Estimated); Last update posted 2011-03-28 (Estimated); Status verified 2011-03

CONDITIONS: Dystonia; Parkinson Disease
MeSH Terms: conditions — Dystonia; Parkinson Disease

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Parkinsonian patients presenting of the dystonia: 15 Parkinsonian patients presenting of the dystonia of ONE or OFF at the time of the phases of driving fluctuations. These patients must present a dystonia of the upper limb, mainly localised than the level of the segment brachial or in distality.
  Interventions: Other: EMG and Kinematics recording
- patients carrying a primary education dystonia affecting: 15 patients carrying a primary education dystonia affecting at least one of the two upper limbs, without excessive involuntary movements
  Interventions: Other: EMG and Kinematics recording
- patients carrying a secondary dystonia: 15 patients carrying a secondary dystonia (consecutive with a perinatal suffering) affecting at least one of the two upper limbs, without excessive involuntary movements
  Interventions: Other: EMG and Kinematics recording
- pilot subjects: 30 healthy pilot subjects paired in sex, age (± 5 years), dominant laterality and level of schooling (15 subjects paired with the Parkinsonian patients and 15 subjects paired with the patients dystonic

INTERVENTIONS:
Other: EMG and Kinematics recording — The experimental protocol envisages the recording of the movement and the bilateral recording of activity EMG during three types of tasks:
  discrete driving tasks: movements of inflection and extension of the wrist car-generated, or produced in answer to an imperative stimulus try driving repetitive: sequence of inflection-extension of the wrist unilateral, bilateral in phase and bilateral in opposition of phase.
  try driving complexes: movement of inflection and extension of the wrist with concurrent realization of a driving task controlatérale different, or of a cognitive task.
  For the Parkinsonian patients, these various tests will be carried out twice: without antiparkinsonian treatment ("off") and under treatment ("one").
  Groups: Parkinsonian patients presenting of the dystonia; patients carrying a primary education dystonia affecting; patients carrying a secondary dystonia

SUMMARY:
Dystonia is a rare disease leading to a severe handicap. It can be of primary or secondary origin. It is characterized by sustained muscle contractions, frequently causing twisting and repetitive movements or abnormal postures. These disorders are believed to be caused by some dysfunction of the basal ganglia (BG) circuitry, but the mechanisms are largely unknown.

A better understanding of the disorder requires significant improvements of its phenomenological description in relation to aetiology. We want to identify specific motor signatures of different forms of dystonia. To that aim, we will ask patients to perform movements of various complexities, while recording chronometric, kinematics and EMG data. The characteristics of the patients' movements will be compared to those of matched control subjects. We will examine abnormal co-activation in distal and proximal muscles to evaluate the characteristics of the loss of selectivity of the motor command in mobile vs. fixed dystonia. Consistency of the motor output patterns will be compared in three groups of patients. We will also study possible cognitive and limbic components of the disease, examining the influence of cognitive and emotional loads on movement production. Eventually we want to refine the criteria used to classify different forms of the disease, thus enabling clinicians to better predict the likely outcome of particular therapeutic procedures.

DETAILED DESCRIPTION:
A major difficulty hindering progress in our understanding of dystonia is the fact that accurate descriptions of the motor signs associated with different forms of the disease are presently lacking. Indeed, different forms of the disease yield symptoms that cannot be distinguished on the basis of current clinical evaluations. We hypothesize that the multiple pathophysiological mechanisms that appear to underlie the motor symptoms of dystonia should induce somewhat different behavioural expressions of the disease, and should also respond differently to deep brain stimulation. As proximal muscles are involved in postural limb stabilisation, we propose to not only study distal, but also proximal and contra-lateral diffusion of the motor command. Our hypothesis is that movement and EMG patterns should diverge depending on the aetiology of the disease and task conditions. In other words, we expect to identify kinematics and EMG signatures specific to different forms of dystonia.

One first step towards improving our knowledge of dystonia is thus to scrutinize the motor output at the behavioural level, relating abnormal movement patterns to specific aetiologies of the disease. Thus, three groups of patients presenting a dystonia of known aetiology (ON and OFF dystonia of Parkinson Disease, Primary dystonia, Secondary dystonia) will be included in the study, as well as two groups of age-matched control subjects.

The first step of our experimental approach will consist in studying the kinematics and EMG patterns of movements performed by the different groups of patients. For studying motor control of the upper limb, we will ask the patients to perform both wrist movements in isolation, or in association with a superimposed motor, cognitive or emotional task. The organisation and abnormalities of movements of the lower limb will be studied following the same rationale, whenever possible. Because of the occurrence of involuntary movements in many patients with dystonia, all behavioural recordings will be performed using telemetric equipment. This will guarantee that patients will not pull off the captors, nor run any risk of getting hurt during the recording sessions.

The measures will include reaction and movement times, as well as the angular displacements of the relevant joints and the bilateral EMG activity of the distal and proximal muscles of the limbs. The spatio-temporal characteristics of the patients' movements will be analyzed using the recorded chronometric, kinematics and EMG data, and compared to those of age-matched control subjects. Muscle activity and movement will be recorded at the different levels of the moving and contralateral limbs to thoroughly monitor of the overflow characteristics of dystonia.

Dystonic bradykinesia is thought to be related to a loss of the selectivity of the motor command, and in particular its diffusion to antagonist groups. If this hypothesis is correct, we expect to observe abnormal co-activation of antagonist groups at the distal level. Because of the postural component of dystonia, we also expect to see an undue diffusion of the motor command to proximal muscles. Finally, we will look for signs of mirror movements indicating perturbations of inter-hemispheric motor inhibition.

The abnormal co-activation of antagonists and proximal muscles should increase under double motor task conditions, where the patient will be asked to perform symmetrical or different movements simultaneously with the two limbs. Based on the hypothesis that symmetrical coupling of motor effectors is easier to control than asymmetrical patterns, which require inter-hemispheric inhibition of the irrelevant movement, motor performance should be more difficult and diffusion of the motor command should be increased in the asymmetrical motor tasks.

Under each condition of movement, the consistency of the recorded patterns of kinematics and EMG data will be compared between the three groups of patients. Regarding secondary dystonia, whenever relevant, we will also correlate the observed patterns with existing cerebral lesions. We will attempt to find further connections between the clinical phenotype of the patients and the measured movement parameters. For example, the kinematics and EMG data will be put into relation to the main types of symptoms displayed by the patients (mobile vs. fixed dystonia), and the distribution of the symptoms.

The hypothesis that dystonia is a pure motor disease will be tested using double task experimental protocols. Patients will be requested to perform the same arm movement, while 1) performing a simultaneous cognitive task, such as counting backwards or detecting a specific visual stimulus, diverting some of the attentional resources.

ELIGIBILITY:
Inclusion Criteria:

* Parkinsonian patients: idiopathic PD, aged 18 to 75 years, with medical insurance, presenting motor fluctuations with ON and OFF involuntary movements, able to sign informed consent, able to stay in a sitting position and perform the experimental tasks.
* Dystonia patients: aged 18 to 75 years, with medical insurance, idiopathic or secondary dystonia affecting at least one of the upper limbs, able to sign informed consent, able to stay in a sitting position and perform the experimental tasks.

Exclusion Criteria:

* Major depression, Dementia, Acute psychosis, Clinical motor deficit making the movements impossible, joint or muscle pathology.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Parkinsonian patients, Dystonia patients,Major depression, Dementia, Acute psychosis, Clinical motor deficit making the movements impossible, joint or muscle pathology
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2006-08; Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bettina DEBU, Professor, Study Director — University J Fourier, INSERM U 318; Pierre POLLAK, Professor, Principal Investigator — University J Fourier, INSERM U318, Grenoble University Hospital
Locations (1):
- Grenoble University Hospital, Grenoble, France